CLINICAL TRIAL: NCT01275157
Title: Disposition of [14C]-LY2452473 Following Oral Administration in Healthy Human Subjects
Brief Title: Disposition of 14C-LY2452473 Following Oral Administration in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13276; I2N-MC-GPBF (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Healthy Volunteers
Keywords: Absorption; Distribution; Metabolism; Excretion; Mass balance; Metabolic profile; Radiolabeled study; 14C
MeSH Terms: interventions — LY2452473

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2452473 (Experimental): 15 mg, containing 100 micro curies of 14C labeled LY2452473 taken once only
  Interventions: Drug: LY2452473

INTERVENTIONS:
Drug: LY2452473 — Administered orally as a liquid suspension

SUMMARY:
This is a single dose study of radiolabeled [14C]-LY2452473 in healthy male volunteers to study the absorption, distribution, metabolism, and elimination of LY2452473.

This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Experience on average 1 to 2 bowel movements per day
* Overtly healthy males, as determined by medical history and physical examination
* Subjects will either be sterile or, if sexually active, agree to use a reliable method of birth control from check-in until 3 months after the follow-up assessment
* Are between the body mass index (BMI) of 19 and 29 kg^m2, inclusive
* Clinical laboratory test results within the normal reference range for the clinical research unit laboratory or results with acceptable deviations which are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow blood sampling
* Normal blood pressure and pulse rate (sitting) as determined by the investigator
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the Institutional Review Board (IRB) governing the site

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device other than the study drug used in this study, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2452473 or related compounds
* Within 30 days of the initial dose of study drug, have received treatment with a drug that has not received regulatory approval for any indication
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study medication or interfering with the interpretation of data
* Have any other condition that in the opinion of the investigator would preclude participation in the study
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Intended use of over-the-counter or herbal medication within 7 days or prescription medication within 14 days prior to dosing
* Have donated more than 500 mL of blood within the last month
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption for the duration of the study (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Use of herbal preparations containing St. John's Wort, kava, garlic, ginger, gingko biloba, or guarana within 14 days prior to admission
* Consumption of grapefruit or grapefruit-containing foods or juices within 7 days prior to dosing or any time during the study
* Heavy caffeine drinkers defined by a regular intake of more than 5 cups (40-50 mg of caffeine per cup) of coffee (or equivalent in xanthine-containing beverages) per day or caffeine drinking subjects who have not had consistent daily caffeine consumption for 1 month prior to study entry or subjects not willing to maintain consistent caffeine consumption during the study
* Have participated in a [14C]-study within the last 12 months. The previous radiolabeled study drug must have been received more than 6 months prior to Check-in for this study and the cumulative annual radiation exposure must be consistent with Food and Drug Administration (FDA) recommendations, for example whole body exposure less than 5,000 mrem/year
* Exposure to significant radiation within 12 months prior to dose (for example, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Urinary and fecal excretion of radioactivity over time expressed as a percentage of the total radioactive dose administered | baseline up to 22 days

SECONDARY OUTCOMES:
Plasma pharmacokinetics of LY2452473 and radioactivity maximum observed concentration (Cmax) | baseline up to 22 days
Plasma pharmacokinetics of LY2452473 and radioactivity time of maximum observed concentration (tmax) | baseline up to 22 days
Plasma pharmacokinetics of LY2452473 and radioactivity area under the concentration-time curve from time zero to the last timepoint with a measurable concentration (AUC 0 to tlast) | baseline up to 22 days
Relative abundance of LY2452473 and the metabolites of LY2452473 in urine and feces | baseline up to 22 days
Relative abundance of LY2452473 and the metabolites of LY2452473 in plasma | baseline up to 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States